CLINICAL TRIAL: NCT02496455
Title: The Impact of the Single Nucleotide Polymorphisms rs6746030,rs7604448, rs10930214, s7595255 in SCN9A Gene on Postoperative Pain and Analgesic Consumption After Cesarean Section
Brief Title: The Impact of the SCN9A Gene Polymorphism on Postoperative Pain
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Tuğba Karaman, Assistant Professor, M.D., Tokat Gaziosmanpasa University
Other Study IDs: GEN-S
Record Dates: First submitted 2015-07-09; First posted 2015-07-14 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-08

CONDITIONS: Pain, Postoperative; Pregnancy
Keywords: NAV1.7 Voltage-Gated Sodium Channel; pain, postoperative; cesarean section
MeSH Terms: conditions — Pain, Postoperative | interventions — Cesarean Section; Tramadol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two ml blood will be collected from the peripheral venous before the operation and all blood samples will be stored at -80℃. Genomic DNA will be extracted from the blood samples and polymorphism in SCN9A gene will be identified by PCR
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: cesarean section — Women in 36 to 40 weeks of pregnancy undergoing cesarean section by Pfannenstiel technique
Drug: Opioid Tramadol — Tramadol will be administered via patient controlled analgesia (PCA) pump in the postoperative period
  Other Names: Tramadol (contramal)

SUMMARY:
The purpose of this study to determine the association between postoperative pain after cesarean section and several single nucleotide polymorphisms in SCN9A sodium channels gene.

DETAILED DESCRIPTION:
SCN9A gene encodes an alpha subunit of the voltage-gated sodium channel (Nav1.7) and polymorphisms of this gene are associated with severe pain disorders. The impact of the polymorphisms in SCN9A on postoperative pain and opioid consumption after cesarean section is unclear.

ELIGIBILITY:
Inclusion Criteria:

* The women aged 18 to 45,
* in 36 to 40 weeks of pregnancy
* undergoing cesarean section

Exclusion Criteria:

* History of chronic pain or pain disorders
* Psychiatric diseases
* Diabetes mellitus
* Severe cardiovascular, kidney or liver diseases
* Alcohol or drug abuse
* Heavy smoker
* Unable to use the Patient controlled analgesia (PCA) pump

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The women in 36 to 40 weeks of pregnancy undergoing cesarean section will be included
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-08; Primary Completion 2017-05 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Pain | up to postoperative 24 hours
  The pain will be evaluated with the visual analog scale

SECONDARY OUTCOMES:
Opioid consumption | Up to postoperative 24 hours
  The total amount of the tramadol administered to the patient will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Karaman, M.D., Principal Investigator — Gaziosmanpasa University Medical School
Locations (1):
- Gaziosmanpasa University Medical School Hospital, Tokat Province, Turkey (Türkiye)